CLINICAL TRIAL: NCT02653534
Title: Impact of Promoting Community Initiated Kangaroo Mother Care (KMC) for Low Birth Weight Infants
Acronym: KMC-LBW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: Centre For International Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/1486/REK vest
Record Dates: First submitted 2015-12-26; First posted 2016-01-12 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2015-12

CONDITIONS: Low-Birth-Weight
Keywords: Kangaroo Mother Care in community; mortality
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Kangaroo Mother Care (Experimental): Promotion of, and support for lactation management and skin to skin care as soon as possible after birth by study ANM supported by study ASHA in addition to routine visits by government health workers
  Interventions: Behavioral: Kangaroo Mother Care
- Control (No Intervention): Routine visits by government health workers

INTERVENTIONS:
Behavioral: Kangaroo Mother Care — Promotion of, and support for lactation management and skin to skin care as soon as possible after birth by study ANM supported by study ASHA in addition to routine visits by government health workers
  Arms: Intervention Kangaroo Mother Care

SUMMARY:
This study is being conducted to assess the impact of promoting community initiated Kangaroo Mother Care (ciKMC) for low birth weight babies on post enrolment neonatal mortality and mortality post enrolment upto 6 months of age. This large individually randomized controlled trial will enroll 10500 low birth weight babies. The secondary objectives are examining the impact of the intervention on exclusive breast feeding and growth at 1 and 3 months, infections and hospitalizations in the neonatal period and from 1 to 5 months of age, recognition of illnesses and early care seeking from appropriate sources, motor and mental development in a subsample.

Newborns weighing >=1500 to <=2250gm are being enrolled into the study within 3 days of birth. Eligible babies are randomized to intervention or control arms. Mothers in the intervention arm are supported for KMC and breastfeeding by study ANM (Auxiliary Nurse Midwife) and study ASHA (Accredited Social Health Activist) like workers . Routine home visits are conducted in both intervention and control arms by government workers according to the existing government program.

Survival will be ascertained in all enrolled infants through contacts at 1, 3 and 6 months.

The data safety and monitoring committee (DSMC) conducted two interim analyses, first in September 2017 when about half of the infants had been enrolled, and second in June 2018, when almost three quarters of the enrolled babies had been followed till 28 days of age. Following the second interim analysis, the DSMC concluded that a sufficient number of infants would be enrolled by the end to September 2018 to clearly answer the study question concerning the impact of ciKMC on both neonatal and early infant mortality. The DSMC recommended that data collection be completed by the end of October 2018.

ELIGIBILITY:
Inclusion Criteria:

Low birth weight babies (≥1500 to ≤2250 g) screened within 3 days and their mothers.

* Born at home
* Singleton or twins or triplets
* Infants born in hospital, discharged and KMC not initiated in the hospital

Exclusion Criteria:

* Infant unable to feed
* Infant has breathing problem
* Infant is less active than normal
* Gross congenital malformations
* Mother does not intend to stay in the study area for the next 6 months

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8402 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Neonatal mortality from post enrolment to 28 days | From post enrolment to 28 days
Early infant mortality from post enrolment to 6 months of age | From post enrolment to 6 months

SECONDARY OUTCOMES:
Proportion exclusively breastfed at 1 and 3 months | 1 month, 3 months
Weight gain | 1, 3 and 6 months
Length gain | 1, 3 and 6 months
Incidence of infection and hospitalization | 1 month and 1 to 5 months
Early recognition of illness at 1 month | 1 month period
  Recognition of illness will be ascertained from caregivers by using questionnaire
Early appropriate care seeking practices at 1 month | 1 month period
  Early appropriate care seeking ascertained from caregivers by using questionnaire
Early recognition of illness at 3 months | Assessed at 3 months, data from 1 month upto 3 months
  Recognition of illness ascertained from caregivers by using questionnaire
Early appropriate care seeking practices at 3 months | Assessed at 3 months, data from 1 month upto 3 months
  Early appropriate care-seeking ascertained from caregivers by using questionnaire
Early recognition of illness at 6 months | Assessed at 6 months, data from 3 months upto 6 months
  Recognition of illness ascertained from caregivers by using questionnaire
Early appropriate care seeking practices at 6 months | Assessed at 6 months, data from 3 months upto 6 months
  Early appropriate care-seeking practices ascertained by using questionnaire
Assessment of cognitive function by Bayley scale in a subsample | Assessment of cognitive function by Bayley scale at 6 months
Assessment of cognitive function by Bayley scale in a subsample | Assessment of cognitive function by Bayley scale at 12 months
Head circumference | 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sarmila Mazumder, MBBS, PhD, Principal Investigator — Society for Applied Studies
Locations (1):
- CHRD, Society for Applied Studies, Palwal, Haryana, India

REFERENCES:
- [Derived] Choudhary TS, Kumar M, Sinha B, Shaikh S, Mazumder S, Taneja S, Bhandari N. Anthropometric Indicators as Predictors of Mortality in Early Life Among Low Birthweight Indian Infants. Front Nutr. 2022 Jul 12;9:884207. doi: 10.3389/fnut.2022.884207. eCollection 2022. PMID 35903458
- [Derived] Sinha B, Choudhary TS, Nitika N, Kumar M, Mazumder S, Taneja S, Bhandari N. Linear Growth Trajectories, Catch-up Growth, and Its Predictors Among North Indian Small-for-Gestational Age Low Birthweight Infants: A Secondary Data Analysis. Front Nutr. 2022 May 24;9:827589. doi: 10.3389/fnut.2022.827589. eCollection 2022. PMID 35685868
- [Derived] Choudhary TS, Mazumder S, Haaland OA, Taneja S, Bahl R, Martines J, Bhan MK, Johansson KA, Sommerfelt H, Bhandari N, Norheim OF. Health equity impact of community-initiated kangaroo mother care: a randomized controlled trial. Int J Equity Health. 2021 Dec 24;20(1):263. doi: 10.1186/s12939-021-01605-0. PMID 34952592
- [Derived] Mazumder S, Taneja S, Dube B, Bhatia K, Ghosh R, Shekhar M, Sinha B, Bahl R, Martines J, Bhan MK, Sommerfelt H, Bhandari N. Effect of community-initiated kangaroo mother care on survival of infants with low birthweight: a randomised controlled trial. Lancet. 2019 Nov 9;394(10210):1724-1736. doi: 10.1016/S0140-6736(19)32223-8. Epub 2019 Oct 4. PMID 31590989
- [Derived] Mazumder S, Taneja S, Dalpath SK, Gupta R, Dube B, Sinha B, Bhatia K, Yoshida S, Norheim OF, Bahl R, Sommerfelt H, Bhandari N, Martines J. Impact of community-initiated Kangaroo Mother Care on survival of low birth weight infants: study protocol for a randomized controlled trial. Trials. 2017 Jun 7;18(1):262. doi: 10.1186/s13063-017-1991-7. PMID 28592313